CLINICAL TRIAL: NCT04681144
Title: Describing the Quality Of Life in Colombian Patients mCRPC Under Treatment With RADium-223.
Brief Title: A Study to Learn More About How Radium-223 Affects the Quality of Life of Colombian Patients With Prostate Cancer That Has Not Responded to Testosterone Lowering Treatment and Has Spread to the Bones, and to Better Understand Its Safety
Acronym: QOLRAD
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21517
Record Dates: First submitted 2020-12-04; First posted 2020-12-23 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-08

CONDITIONS: Prostate Cancer
Keywords: Bone metastatic castration resistant prostate cancer; Radium-223; mCRPC; Phase IV; Advance prostate cancer; Quality of life; Bone Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Bone Neoplasms | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radium-223-dichloride (Xofigo, BAY88-8223): Patients with metastatic castration-resistant prostate cancer (mCRPC)
  Interventions: Drug: Radium-223-dichloride (Xofigo, BAY88-8223)

INTERVENTIONS:
Drug: Radium-223-dichloride (Xofigo, BAY88-8223) — Decision to initiate treatment with Radium-223 made as per investigator's routine treatment practice

SUMMARY:
The study drug, radium-223, gives off radiation that helps to kill cancer cells in the prostate. It is already available for patients to receive as a treatment for prostate cancer that has not responded to testosterone lowering treatment and has spread to the bones. This type of cancer is called metastatic castration-resistant prostate cancer, also called mCRPC. Sometimes, researchers continue studying an available treatment to learn more about how it affects patients' daily lives.

In this study, the researchers want to learn more about how radium-223 affects the patients' ability to do their daily tasks. The patients in this study will already be receiving treatment with radium-223 as part of their routine care. The tests and measurements in this study will be done by the patients' own doctors. The researchers will collect information about the patients' treatment and results.

The study will include patients with mCRPC who have at least 2 tumors in their bones. These patients will have recently started treatment with radium-223. The patients will have also had surgery or treatment to lower their testosterone levels. But, the treatment did not help their cancer. The study will include about 105 men in Colombia who are at least 18 years old.

All of the patients will receive radium-223 through a needle put into the vein, also called an intravenous injection. They will visit their doctor's office up to 8 times during 28 weeks. At these visits, their doctors will ask how they are feeling and what medications they are taking, and will take blood samples. The doctors will also give the patients surveys about their physical, social, and emotional health and about the symptoms of their prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male adult patients (> 18 years)
* Label Xofigo
* Signed informed consent
* No participation in an investigational program with interventions outside of routine clinical practice.
* Decision to initiate treatment with Radium-223 made as per investigator's routine treatment practice, as treatment option for mCRPC either as first line (naïve), second line (after progression during treatment with enzalutamide or abiraterone) or third line (post-Docetaxel).

Exclusion Criteria:

* Patients with contraindications to the use of Radium-223 according to the local label.
* Patients and who refused to sign the informed consent form.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colombian patients diagnosed with metastatic castration-resistant prostate cancer (mCRPC).
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Absolute scores for FACT-P | At baseline
  Functional Assessment of Cancer Therapy-Prostate (FACT-P): It is a multidimension, selfreport QoL instrument specifically designed for patients with prostate cancer. It consists of 39 questions items, made up by 2 parts: the 27 questions for functional assessment of cancer therapy general (FACT-G) and 12 prostate cancer subscale questions. It assesses 4 main domains which are: physical (n=7), social/family (n=7), emotional (n=6) and functional wellbeing (n=7).
Absolute scores for FACT-P | At week 12
Absolute scores for FACT-P | At week 16
Absolute scores for FACT-P | At week 24
Absolute scores for FACT-P | At week 28
Absolute scores for EORTC QLQ-PR25 | At baseline
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Prostate Specific module (EORTC QLQ-PR25): It is a questionnaire with score calculation is by subscales: urinary symptoms, bother due to use of incontinence aid, bowel symptoms, hormonal treatment-related symptoms, sexual activity and sexual functioning. Absolute score [scores are linearly transformed to a 0-100 scale, with higher scores reflecting either more symptoms (urinary, bowel, hormonal treatment-related symptoms) or higher levels of activity or functioning (sexual).
Absolute scores for EORTC QLQ-PR25 | At week 12
Absolute scores for EORTC QLQ-PR25 | At week 16
Absolute scores for EORTC QLQ-PR25 | At week 24
Absolute scores for EORTC QLQ-PR25 | At week 28

SECONDARY OUTCOMES:
Absolute scores for Physical Well Being, Social/Family Well Being, Emotional Well Functional Well Being, in the FACT-P | Baseline, 12, 16, 24- and 28-weeks and follow up visit week 28; 4 weeks post last injection
Absolute scores for urinary and bowel symptoms, sexual activity and function, and adverse effects to treatments in the EORTC QLQ-PR25 | Baseline, 12, 16, 24- and 28-weeks and follow up visit week 28; 4 weeks post last injection
Absolute scores for FACT-P; according to number of Radium-223 cycles | Baseline, 12, 16, 24- and 28-weeks and follow up visit week 28; 4 weeks post last injection
  Number of cycles of Radium-223 will be measured as total number of doses received.
Absolute scores for EORTC QLQ-PR25; according to number of Radium-223 cycles | Baseline, 12, 16, 24- and 28-weeks and follow up visit week 28; 4 weeks post last injection
  Number of cycles of Radium-223 will be measured as total number of doses received.
Absolute scores for FACT-P; according line of treatment | Baseline, 12, 16, 24- and 28-weeks and follow up visit week 28; 4 weeks post last injection
  Line of treatment is classified as first , second or third line agent according to formulation scheme.
Absolute scores for EORTC QLQ-PR25; according line of treatment | Baseline, 12, 16, 24- and 28-weeks and follow up visit week 28; 4 weeks post last injection
  Line of treatment is classified as first , second or third line agent according to formulation scheme.
Absolute scores for FACT-P; according to prior use or chemotherapy | Baseline, 12, 16, 24- and 28-weeks and follow up visit week 28; 4 weeks post last injection
  Patients will be classified as prior chemotherapy or chemotherapy naïve
Absolute scores for EORTC QLQ-PR25; according to prior use or chemotherapy. | Baseline, 12, 16, 24- and 28-weeks and follow up visit week 28; 4 weeks post last injection
  Patients will be classified as prior chemotherapy or chemotherapy naïve
Absolute scores for FACT-P; according to clinical characteristics. | Baseline, 12, 16, 24- and 28-weeks and follow up visit week 28; 4 weeks post last injection
  Clinical characteristics: Eastern Cooperative Oncology Group (ECOG) 0-1, more than 2 bone metastasis, no visceral metastasis, Neutrophils: > 1.500 L (>1.5 x10exp9/L, Hemoglobin: > a 10 g/dL, Platelets: > a 100.000 (>100x10exp9/L).
Absolute scores for EORTC QLQ-PR25; according to clinical characteristics. | Baseline, 12, 16, 24- and 28-weeks and follow up visit week 28; 4 weeks post last injection
  Clinical characteristics: ECOG 0-1, more than 2 bone metastasis, no visceral metastasis, Neutrophils: > 1.500 L (>1.5 x10exp9/L, Hemoglobin: > a 10 g/dL, Platelets: > a 100.000 (>100x10exp9/L).
Absolute scores for FACT-P; according to changes in PSA. | Baseline, 12, 16, 24- and 28-weeks and follow up visit week 28; 4 weeks post last injection
  Prostate specific antigen (PSA) level will be measured in subject's blood from baseline and every 2 months after that in accordance with the San Gallen protocol(3) stablish in the routine clinical practice as guidelines for management. The percent change from the baseline value will be calculated as followed: (PSA level at week n - PSA level from baseline)/(PSA level from baseline)*100
Absolute scores for EORTC QLQ-PR25; according to changes in PSA | Baseline, 12, 16, 24- and 28-weeks and follow up visit week 28; 4 weeks post last injection
  PSA level will be measured in subject's blood from baseline and every 2 months after that in accordance with the San Gallen protocol(3) stablish in the routine clinical practice as guidelines for management. The percent change from the baseline value will be calculated as followed: (PSA level at week n - PSA level from baseline)/(PSA level from baseline)*100
Absolute scores for FACT-P; according to changes in ALP level | Baseline, 12, 16, 24- and 28-weeks and follow up visit week 28; 4 weeks post last injection
  Alkaline phosphatase (ALP) level will be measured in subject's blood from baseline and every 2 months after that in accordance with the San Gallen protocol(3) stablish in the routine clinical practice as guidelines for management. The percent change from the baseline value will be calculated as followed: (ALP level at week n - ALP level from baseline)/(ALP level from baseline)*100
Absolute scores for EORTC QLQ-PR25; according to changes in ALP level | Baseline, 12, 16, 24- and 28-weeks and follow up visit week 28; 4 weeks post last injection
  ALP level will be measured in subject's blood from baseline and every 2 months after that in accordance with the San Gallen protocol(3) stablish in the routine clinical practice as guidelines for management. The percent change from the baseline value will be calculated as followed: (ALP level at week n - ALP level from baseline)/(ALP level from baseline)*100

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Colombia

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.